CLINICAL TRIAL: NCT03376802
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Repeated Subcutaneous Doses of SAR425899 on Energy Expenditure and Safety in Overweight to Obese Male and Female Subjects
Brief Title: A Clinical Study to Investigate the Effect of SAR425899 on Energy Expenditure in Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PDY15012; U1111-1191-5658 (Other: UTN)
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR425899

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SAR425899 (Experimental): Repeated once daily subcutaneous (SC) doses of SAR425899 administered over 19 days
  Interventions: Drug: SAR425899
- Placebo (Placebo Comparator): Repeated once daily SC doses of placebo administered over 19 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR425899 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: SAR425899
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess in overweight to obese subjects the change in sleep energy expenditure after repeated subcutaneous (SC) doses of SAR425899.

Secondary Objectives:

* To assess the change in resting, basal and total daily energy expenditure.
* To assess the change in respiratory quotient, fat, protein and carbohydrate oxidation.
* To assess the change in body composition and core temperature.
* To assess the pharmacodynamic effects on fasting plasma glucose, biomarkers of lipid metabolism and glycated hemoglobin (HbA1c).
* To assess the pharmacokinetic parameters for SAR425899 after repeated SC doses.
* To assess the safety and tolerability.

DETAILED DESCRIPTION:
Study duration is approximately 7-8 weeks including a screening period, a 19-day treatment period and an end-of-study visit 7 days after last dosing.

ELIGIBILITY:
Inclusion criteria:

* Overweight to obese male and female subjects.
* Body mass index 28 - 40 kg/m2.
* 18 to 50 years of age
* Fasting plasma glucose ≤125 mg/dL.
* Glycated hemoglobine (HbA1c) ≤6.5%.
* Obesity associated mild concomitant diseases allowed (eg, mild hypertension, mild hypercholesteremia, and hyperlipidemia).
* No concomitant medication allowed except stable treatment with statins or antihypertensive drugs (except ß-blocker).
* Females should be either postmenopausal, or, if perimenopausal should have a normal regular menstrual cycle and should start or continue stable treatment with a monophasic oral contraceptive.

Exclusion criteria:

* Elevated liver enzymes, lipase, amylase, or calcitonin at screening.
* Current participation in an organized diet / weight reduction program or clinical trial of weight control or weight loss attempt, plans for major changes in physical activities or significant change in body weight in the 2 months prior to screening.
* Any condition possibly affecting gastric emptying or absorption from gastro-intestinal tract (eg, gastric surgery, gastrectomy, bariatric surgery, malabsorption syndromes, gastroparesis, abdominal surgery other than appendectomy or hysterectomy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Sleep energy expenditure | Baseline to Day 19
  Change of sleep energy expenditure from baseline to Day 19 with SAR425899 or placebo

SECONDARY OUTCOMES:
Total daily energy expenditure | Baseline to Day 19
  Change of total energy expenditure from baseline to Day 19 with SAR425899 or placebo
Resting energy expenditure | Baseline to Day 19
  Change of resting energy expenditure from baseline to Day 19 with SAR425899 or placebo
Basal energy expenditure | Baseline to Day 19
  Change of basal energy expenditure from baseline to Day 19 with SAR425899 or placebo
Respiratory quotient (RQ) | Baseline to Day 19
  Change of respiratory quotient from baseline to Day 19 with SAR425899 or placebo
Fat mass and fat-free mass | Baseline to Day 20
  Change of fat mass and fat-free mass by dual energy X-ray absorptiometry (DEXA) scan from baseline to Day 20 with SAR425899 or placebo
Diet Induced Thermogenesis (DIT) | Baseline to Day 19
  Change of DIT from baseline to Day 19 with SAR425899 or placebo
Fasting plasma glucose | 20 days
  Change of FPG over time with SAR425899 or placebo
HbA1c | Baseline to Day 20
  Change of HbA1c from baseline to Day 20 with SAR425899 or placebo
Lipid biomarker (free fatty acids, triglycerides, total cholesterol, HDL-/LDL-cholesterol) | 20 days
  Change of lipid biomarkers over time with SAR425899 or placebo
Ketone bodies | 20 days
  Change of ketone bodies over time with SAR425899 or placebo
Adverse events | Up to 27 days
  Number of adverse events in patients under treatment with SAR425899 or placebo
Pharmacokinetics | Day 16
  Assessment of SAR425899: time to reach Cmax (tmax)
Pharmacokinetics | Day 16
  Assessment of SAR425899: maximum plasma concentration (Cmax)
Pharmacokinetics | Day 16
  Assessment of SAR425899: area under the concentration versus time curve (AUC)
Pharmacokinetics | Day 16
  Assessment of SAR425899: terminal elimination half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number 8400001, Orlando, Florida
  - Investigational Site Number 8400002, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org